CLINICAL TRIAL: NCT05414123
Title: A Longitudinal Therapy Response Monitoring Study in Subjects With Leptomeningeal Metastases Using CNSide (CSF Tumor Cells) Compared to Standard of Care (CSF Cytology, Clinical Evaluation, and Imaging).
Brief Title: A Therapy Treatment Response Trial in Patients With Leptomeningeal Metastases ((LM) Using CNSide
Acronym: FORESEE
Status: Terminated | Type: Observational
Why Stopped: The sponsor can no longer financially support the trial.
Sponsor: Biocept, Inc. (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Other Study IDs: BIOC-046
Record Dates: First submitted 2022-06-08; First posted 2022-06-10 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Leptomeningeal Metastasis; Leptomeningeal Disease; Leptomeningeal Neoplasms; Breast Cancer; Non-Small Cell Lung Cancer
Keywords: Leptomeningeal Metastasis; Cerebro-Spinal Fluid; Liquid Biopsy; Tumor Cells
MeSH Terms: conditions — Meningeal Carcinomatosis; Meningeal Neoplasms; Breast Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Breast Cancer: Subjects with Breast Cancer of all subtypes and independent of Hormone status who have a confirmed or suspicious Leptomeningeal Metastasis by Investigator assessment of radiographic image and clinical evaluation and cytology
  Interventions: Device: CNSide
- Non-Small Cell Lung Cancer: Subjects with Non-Small Cell Lung Cancer of all subtypes who have a confirmed or suspicious Leptomeningeal Metastasis by Investigator assessment of radiographic image and clinical evaluation and cytology
  Interventions: Device: CNSide

INTERVENTIONS:
Device: CNSide — The Cerebro-Spinal Fluid (CSF) of subjects enrolled into each cohort will be used for Standard of Care diagnostic assessments used for subjects with either confirmed or suspicious LM (Cytology, protein and glucose) in combination with CNSide analysis.

SUMMARY:
The FORESEE Study is a multi-center, prospective clinical trial enrolling patients with Breast or Non-Small Cell Lung Cancer (NSCLC) who have suspicious or confirmed Leptomeningeal Metastases (LM). Standard of Care methods to diagnose, or assess the treatment response of LM (Clinical Evaluation, MRI and Cytology) have limited sensitivity and specificity. This creates challenges for physicians to manage LM or determine the best course of treatment. CNSide, is a Laboratory Developed Test (LDT ) that is used commercially at the Physician's discretion in Biocept's CLIA certified, CAP accredited laboratory. CNSide can detect and quantify tumor cells in the CSF from patients with Breast Cancer or NSCLC having a suspicious or confirmed LM. The goal of the FORESEE Study is to evaluate the performance of CNSide in monitoring the LM's response to treatment and to assess the impact of CNSide on treatment decisions made by Physicians.

DETAILED DESCRIPTION:
The FORESEE Study is a multi-center, prospective clinical trial enrolling patients with breast or Non-Small Cell Lung Cancer (NSCLC) who have suspicious or confirmed Leptomeningeal Metastases (LM). LM is a devastating complication of breast cancer and NSCLC and is diagnosed via clinical evaluation, MRI (with and without contrast of the brain and spine), and CSF Cytology. These methods have limited sensitivity and specificity. Furthermore, they lack the ability to quantitatively measure the LM's response to treatment. These hindrances create challenges for physicians to manage LM or to determine the best course of treatment. CNSide, is a Laboratory Developed Test (LDT ) that is analytically validated and run commercially in Biocept's CLIA certified, CAP accredited laboratory at the Physician's discretion. CNSide can detect and quantify tumor cells in the CSF from patients with Breast Cancer or NSCLC having a suspicious or confirmed LM. Data derived from case studies suggest that the detection of tumor cells in the CSF by CNSide can be used by Physicians to monitor the response of the LM tumor to treatment and improve the ability to make treatment decisions in patients with LM. Subjects enrolled onto the trial will be treated per Standard of Care. The diagnostic tests used to either diagnose LM, or monitor the LMs response to treatment will be Standard of Care, in combination with CNSide. The goal of the FORESEE Study is to further evaluate the performance of CNSide for LM in monitoring the LM's response to treatment and to assess the impact of CNSide on treatment decisions made by Physicians.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects => 18 years of age
2. All genders, races, or ethnic groups,
3. Diagnosed with Breast Cancer or NSCLC who present with clinically suspected LM based on Investigator assessment of radiographic image, cytology, and clinical evaluation.
4. Cytology positive and negative subjects will be included.
5. Subjects willing to provide an Informed Consent.
6. Subjects willing and able to undergo CSF or blood collection via Lumbar Puncture and Ommaya Reservoir as well as veni-puncture and shunt.
7. Both patients with and without parenchymal brain metastases will be eligible as long as leptomeningeal metastases are suspected
8. Subjects who previously had a diagnosis of Leptomeningeal Disease by Investigator assessment of radiographic image and clinical evaluation and cytology.

Exclusion Criteria:

1. Subjects who do not have cancer,
2. Subjects with other types of tumors than breast or lung cancer
3. Subjects diagnosed with a primary brain tumor
4. Subjects who are unable to undergo lumbar puncture, a shunt or veni-puncture.
5. Lack of suspicious LM based in imaging or clinical evaluation.
6. Ordering the Commercial CNSide test while subject is on study
7. Pregnant women and adults lacking capacity to consent for themselves

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subjects will be selected from all clinics where subjects having Breast Cancer or Non-Small Cell Lung Cancer having a suspicious or confirmed LM are being diagnosed or treated by Physicians.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
Assess the impact of CNSide on treatment decisions | 1 year
  The proportion of decision points during LM treatment in which the physician indicated that CNSide aided in their decision making.

SECONDARY OUTCOMES:
Evaluate CNSide as a treatment response monitoring device for LM tumors | 2 years
  The correlation of changes in tumor cell number throughout treatment with clinical evaluation, cytology, and radiographic results.
The performance of CNSide of tumor cell detection in the CSF compared to cytology | 2 years
  The comparison of the sensitivity, specificity, PPV and NPV of CNSide to cytology in detection of tumor cells in the CSF (Cytology being the reference standard)

CONTACTS AND LOCATIONS:
Overall Officials: Priya Kumthekar, MD, Principal Investigator — Northwestern University Medical Center
Locations (4):
- United States (4):
  - Stanford University, Stanford, California
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
There is no plan to make the IDP available to other researchers.